CLINICAL TRIAL: NCT03427190
Title: Assessment of Preventive Efficacy of an Algorithm Taking Place After Suicide Attempts Among Attempters Admitted to Hospital in the French Overseas Territories
Brief Title: Suicide Prevention Algorithm in the French Overseas Territories
Acronym: APSOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Center of Martinique (Other)
Collaborators: Centre Hospitalier de Monteran, Guadeloupe (Unknown); Centre Hospitalier Universitaire de la Guadeloupe (Other); Centre Hospitalier de Cayenne (Other); Centre Hospitalier de Ouest Guyanais Franck Joly (Unknown); Centre d Accueil Psychiatrique Ouest-Centre, La Réunion (Unknown); Centre d Accueil d Urgences Médico Psychologique, La Réunion (Unknown); Centre d Accueil Psychiatrique Nord, La Réunion (Unknown); Etablissement Publique de Santé Mentale de la Réunion (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15/B/04
Record Dates: First submitted 2017-01-30; First posted 2018-02-09 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2020-10

CONDITIONS: Suicide Attempt
Keywords: Suicide; Suicide attempted; Secondary Prevention; Relapse prevention; Case Management; Intervention Study
MeSH Terms: conditions — Suicide, Attempted; Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Phone contact with patient will be made by a professional psychologist within 21 days of hospital discharge. If contact cannot be made after 9 attempts, post-cards will be sent monthly at M2, M3, M4 and M5, asking the participant to establish contact with the designated psychologist. The phone call will determine whether or not the participant is in a state of suicidal crisis. If yes, steps will be taken to attend the crisis within 24 hours.
  Interventions: Other: APSOM vs Control
- APSOM (Other): In complement to actions described in the control arm, the patient's general practitioner (GP) and the patient him/herself will be contacted within 21 days of hospital discharge in order to organize an appointment between them two; this consultation is expected to take place between day 22 and day 45 after hospital discharge. If the patient does not have a GP, a health-care professional (HCP) will be provided. .GP (or HCP) will also be contacted at 6 and 13 months.
  Interventions: Other: APSOM vs Control

INTERVENTIONS:
Other: APSOM vs Control — In complement to actions described in the control arm, the patient's general practitioner (GP) and the patient him/herself will be contacted within 21 days of hospital discharge in order to organize an appointment between them two; this consultation is expected to take place between day 22 and day 45 after hospital discharge. If the patient does not have a GP, a health-care professional (HCP) will be provided. .GP (or HCP) will also be contacted at 6 and 13 months.

SUMMARY:
In France, suicide behaviours are a major public health concern that triggered the creation in 2013 of a National Observatory of Suicide. In continental France, the "Algos" protocol was found to be effective for the prevention of suicide attempts reiterations. This protocol is based on a procedure that keeps telephone and postal contacts with the suicide attempter and allows, via an algorithm, to assess the risk of suicide attempt recurrence, in order to intervene if necessary. Nevertheless, Algos does not involve primary care health practitioners, who could add a substantial additional efficacy, especially if they intervene downstream and in supplement to Algos. In addition, this kind of protocol has never been evaluated in the French overseas territories.

DETAILED DESCRIPTION:
Since (1) Algos was never implemented in the French overseas departments (FOD) and does not involve primary care practitioners (PCP), (2) the additional effect of PCP involvement over and beyond Algos alone in unknown, and (3) little research on suicide behaviours has been conducted in the FOD, this proposal has the following main aim: to assess the effectiveness and the efficacy of the intervention, in supplement and downstream to Algos, of a healthcare professional, on the recurrence of suicide attempts in the FOD; the healthcare professional will be the patient's general practitioner, whenever possible.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman over 16 years of age
* Leaving the hospital within 15 days of the suicide attempt
* Giving (him/herself or his/her legal representative)an oral consent to participate in the study
* Having healthcare insurance
* Reachable by phone, with possibility of confidential conversation, and by mail
* Resident of Guadeloupe, French Guyana, Martinique, or Reunion Island
* Able to understand and speak French

Exclusion Criteria:

* Homeless person
* Disabled adult, person under judicial/court protection, legally incompetent adult
* Participant unable to understand the study protocol, its risks and side effects, or declining to participate

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
Existence of a suicide | 6 months
  Reiteration of suicidal attempt after hospital discharge
Existence of a suicide | 13 months
  Reiteration of suicidal attempt after hospital discharge

SECONDARY OUTCOMES:
Number of suicide attempts | 6 and 13 months after hospital discharge
  To know total number of suicide
Number of deaths by suicide | 6 and 13 months after hospital discharge
  To know number of deaths by suicide
Scores at the Hospital Anxiety and Depression Scale (HADS) | 6 and 13 months after hospital discharge
  Pass the scale HADS
Assessment of suicidal risk by the Sad Persons Scale and the Columbia Suicide Severity Rating Scale (C-SSRS). | 6 and 13 months after hospital discharge
  Pass the scale Columbia

CONTACTS AND LOCATIONS:
Overall Officials: JEHEL Louis, MD-PhD, Principal Investigator — CHU de Martinique
Locations (9):
- French Guiana (2):
  - CH de Cayenne, Cayenne
  - CH Ouest Guyanais, Saint-Laurent-du-Maroni
- Guadeloupe (2):
  - CHU de Pointe à Pitre, Les Abymes
  - CH de Monteran, Saint-Claude
- CHU Martinique, Fort-de-France, Martinique
- Reunion (4):
  - Etablissement Psychiatrique de Santé Mentale, Saint-Benoît
  - Centre d'Accueil Psychiatrique Nord, Saint-Denis
  - Centre d'Accueil Psychiatrique Ouest-Centre, Saint-Paul
  - Centre d'Accueil d'Urgences Médico-Psychologique, Saint-Pierre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617